CLINICAL TRIAL: NCT02379572
Title: Impact of iMRI on the Extent of Resection in Patients With Newly Diagnosed Glioblastomas - A Prospective Multicenter Parallel Group Clinical Trial
Brief Title: Impact of iMRI on the Extent of Resection in Patients With Newly Diagnosed Glioblastomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nch1
Record Dates: First submitted 2015-02-18; First posted 2015-03-05 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2020-07

CONDITIONS: Glioblastoma
Keywords: 5-ALA; Intraoperative MRI; Extent of resection
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- iMRI-guided surgery (Experimental): Resection of Glioblastomas with iMRI-guidance
  Interventions: Device: iMRI-guided surgery
- 5-ALA-guided surgery (Active Comparator): Resection of Glioblastomas with 5-ALA-fluorescence-guidance
  Interventions: Drug: 5-ALA-guided surgery

INTERVENTIONS:
Device: iMRI-guided surgery — For iMRI-guided glioma resections the surgery can be paused and a direct intraoperative resection control is possible by performing an intraoperative MRI scan. If residual tumor is found, the resection might be continued.
  Arms: iMRI-guided surgery
Drug: 5-ALA-guided surgery — For 5-ALA guided glioma resections patients have to drink 100ml of a solution with 5-Aminolevulinic acid 4-6 hours before surgery. Intraoperatively the light source of the surgical microscope can be switched to a certain wave length to enable fluorescence of the glioma cells, which helps resecting the tumor as radical as possible.
  Arms: 5-ALA-guided surgery

SUMMARY:
Standard treatment of glioblastomas (GBMs) consists of microsurgical resection followed by concomitant chemoradiation. The extent of resection is one of the most important prognostic factors with significant influence on the survival of patients. State of the art technique to achieve the most radical resection possible in conventional surgery is fluorescence-guidance with 5-aminolevulinic acid (5-ALA). If available, intraoperative MRI (iMRI)-guided tumor resection enables an intraoperative resection control and subsequent continuation of surgery if contrast enhancing tumor remnants are found. Therefore a more radical resection and longer survival of patients might be possible. To date no comparison of these two leading technologies for GBM-surgery is available to identify the best surgical therapy of this fatal disease and to justify significant healthcare-economic differences between both technologies.

Goal of this study is to assess the value of iMRI guidance in the resection of GBMs in comparison to conventional 5-ALA microsurgery. Primary endpoint is the number of total resections (no residual contrast enhancement) in the postoperative MRI (T1+CM within 48 hours after surgery) in each group. Secondary endpoints are perioperative clinical data, progression free survival, patients' clinical condition and overall survival.

The study design was chosen to be a parallel-group approach to compare iMRI and 5-ALA centers (n=13) to exclude possible bias which might be found by randomizing patients within individual iMRI centers and to have surgeons with the most experience possible in use of each respective technology.

ELIGIBILITY:
Inclusion Criteria:

1. In MRI suspected primary singular untreated GBM
2. Planned total resection of the tumor according to the surgeon
3. Patient ≥18 years, ≤80 years
4. Preoperative KPS ≥ 60%, American Society of Anesthesiologists (ASA) score 1 and 2
5. Patients' informed consent

Exclusion Criteria:

1. Tumors of the midline, basal ganglia, cerebellum, brain stem, eloquent areas
2. Multifocal glioblastoma
3. Substantial (>50%), non-contrast enhancing tumor areas suggesting low-grade glioma with malignant transformation
4. Contraindications to MRI
5. Inability to give consent because of language barrier or dysphasia
6. Histological diagnosis other than Glioblastoma multiforme WHO °IV
7. Increased risk of thrombosis (e.g. Factor V Leiden)
8. Pregnancy or breast feeding
9. Hypersensibility for 5-ALA oder porphyrins
10. Acute or chronic Porphyria
11. Renal insufficiency
12. Hepatic insufficiency
13. High likelihood of inability to receive adjuvant therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2015-06; Primary Completion 2020-06 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Complete resections in the postoperative MRI (T1+/-CM) within 48 hours after surgery | 48 hour
  Completeness of resection in the postoperative MRI within 48h after surgery. Blinded analysis by an independent radiologist.

SECONDARY OUTCOMES:
Patients' clinical condition (KPS) | preoperative (day before surgery), 1 week, 3Months, 6Months, 9Months, 12Months after surgery
  -KPS clinical scoring
Patients' clinical condition (NIHSS) | preoperative (day before surgery), 1 week, 3Months, 6Months, 9Months, 12Months after surgery
  -NIHSS stroke score
Patients' clinical condition (QoL) | preoperative (day before surgery), 1 week, 3Months, 6Months, 9Months, 12Months after surgery
  -quality of life (EORTC) questionnaire
ICU and hospital stay after surgery | Time of hospital stay (average 7days)
  -ICU and overall hospital stay after surgery
Patients' adjuvant treatment | 3Months, 6Months, 9Months, 12Months after surgery
  -adjuvant treatment each patient has received
Recurrent tumor growth (RANO criteria) | 3Months, 6Months, 9Months, 12Months after surgery
  -recurrent tumor growth (RANO criteria) according to local tumor boards and independent blinded analysis
Follow-up imaging | 3Months, 6Months, 9Months, 12Months after surgery
  -follow-up imaging 3, 6, 9, 12 months postoperative incl. independent blinded analysis
Histology | 1 week after surgery
  Histological analysis
MGMT (O6-methylguanine-DNA-methyltransferase) analysis | 1 week after surgery
  MGMT promoter analysis (Routine molecular diagnostics)
IDH-1 (isocitrate dehydrogenase) analysis | 1 week after surgery
  IDH-1 mutation analysis (Routine molecular diagnostics)
Progression-free survival (PFS) | Day of surgery - 6 months - 12 months
  6M&12M-PFS
Overall survival (OS) | Day of surgery - Death of patient (Max. 10 years follow-up)
  OS of patients

OTHER OUTCOMES:
Preoperative tumor localization and resectability concerning eloquent regions | Blinded analysis of preoperative imaging (not older than 3 days prior to surgery)
  Independent blinded analysis of the preoperative imaging data by a blinded neurosurgeon with extensive experience in the resection of gliomas. Analysis will be done before the final evaluation of results. (Within 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Constantin Roder, Dr., Principal Investigator — University Hospital Tuebingen, Department of Neurosurgery
Locations (15):
- Germany (15):
  - Department of Neurosurgery, Universitätsklinikum Bonn, Bonn, Germany, Bonn
  - Department of Neurosurgery, Universität zu Köln, Köln, Germany, Cologne
  - Städtisches Klinikum Dresden Friedrichstadt, Dresden
  - Department of Neurosurgery, Heinrich-Heine-Universität Düsseldorf, Düsseldorf, Düsseldorf
  - Department of Neurosurgery, Friedrich-Alexander-University Erlangen-Nürnberg, Erlangen
  - Department of Neurosurgery, Johann Wolfgang Goethe-University Frankfurt am Main, Frankfurt a.M.
  - Department of Neurosurgery, Georg-August-Universität Göttingen, Göttingen,, Göttingen
  - Department of Neurosurgery, University of Ulm, Hospital Günzburg,, Günzburg
  - Asklepios Klinik Hamburg, Klinik für Neurochirurgie, Hamburg
  - International Neuroscience Institute Hannover, Hannover, Germany, Hanover
  - Department of Neurosurgery, Ruprecht-Karls-University Heidelberg, Heidelberg
  - Department of Neurosurgery, University of Schleswig-Holstein, Kiel, Germany, Kiel
  - Department of Neurosurgery, Westfälische Wilhelms-Universität Münster, Münster, Germany, Münster
  - Department of Neurosurgery, Eberhard Karls University, Tübingen,, Tübingen
  - Department of Neurosurgery, Julius-Maximilians-Universität Würzburg, Würzburg

REFERENCES:
- [Derived] Roder C, Stummer W, Coburger J, Scherer M, Haas P, von der Brelie C, Kamp MA, Lohr M, Hamisch CA, Skardelly M, Scholz T, Schipmann S, Rathert J, Brand CM, Pala A, Ernemann U, Stockhammer F, Gerlach R, Kremer P, Goldbrunner R, Ernestus RI, Sabel M, Rohde V, Tabatabai G, Martus P, Bisdas S, Ganslandt O, Unterberg A, Wirtz CR, Tatagiba M. Intraoperative MRI-Guided Resection Is Not Superior to 5-Aminolevulinic Acid Guidance in Newly Diagnosed Glioblastoma: A Prospective Controlled Multicenter Clinical Trial. J Clin Oncol. 2023 Dec 20;41(36):5512-5523. doi: 10.1200/JCO.22.01862. Epub 2023 Jun 19. PMID 37335962